CLINICAL TRIAL: NCT01902290
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Brodalumab in Subjects With Inadequately Controlled Asthma and High Bronchodilator Reversibility
Brief Title: Study of Efficacy and Safety of Brodalumab Compared With Placebo in Adults With Inadequately Controlled Asthma With High Bronchodilator Reversibility
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to lack of efficacy observed following interim analysis in Q2 2015. Study Closed once all sites were closed in eClinical
Sponsor: Amgen (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120141; 2012-003351-11 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-07-18 (Estimated); Results first posted 2022-02-28 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Asthma
Keywords: Inadequately controlled asthma, brodalumab, AMG 827
MeSH Terms: conditions — Asthma | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo administered by subcutaneous injection on day 1, week 1, week 2 and every 2 weeks thereafter for 24 weeks.
  Interventions: Biological: Placebo
- Brodalumab 210 mg (Experimental): Participants received 210 mg brodalumab administered by subcutaneous injection on day 1, week 1, week 2, and every 2 weeks thereafter for 24 weeks.
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Placebo — Placebo administered subcutaneously
  Arms: Placebo
Biological: Brodalumab — Brodalumab administered subcutaneously
  Other Names: AMG 827
  Arms: Brodalumab 210 mg

SUMMARY:
The purpose of this study is to determine if brodalumab (AMG 827) is safe and effective compared to placebo as measured by change in Asthma Control Questionnaire (ACQ) composite scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, and presently has reversibility over pre-bronchodilator forced expiratory volume in 1 second (FEV1) of ≥ 20% at screening
* Percent of predicted FEV1 ≥ 40% and ≤ 80% at screening
* Inhaled corticosteroid (ICS) ≥ 200 and ≤ 1000/μg/day fluticasone powder or equivalent
* Ongoing asthma symptoms with asthma control questionnaire (ACQ) composite score at screening and baseline ≥ 1.5 points

Exclusion Criteria:

* History of chronic obstructive pulmonary disease (COPD) or other chronic pulmonary condition other than asthma
* History of allergic bronchopulmonary aspergillosis
* Respiratory infection within 4 weeks of screening or 1 week of baseline visit
* Subject has known history of Crohn's disease
* Subject has any other significant concurrent medical condition of laboratory abnormalities, as defined in the study protocol
* Subject has previously used any anti-interleukin-17 (IL17) biologic therapy
* Subject is pregnant or breastfeeding, or planning to become pregnant while enrolled in the study
* Female subject is unwilling to use highly effective methods of birth control unless 2 years post-menopausal or surgically sterile
* Subject has severe depression measured by Personal Health Questionnaire Depression Scale (PHQ-8) or suicidal ideation/behavior as measured by and Columbia Suicide Severity Rating Scale (e-CSSRS)
* Subject has a history or evidence of psychiatric disorder or substance abuse considered by the Investigator to pose a risk to subject safety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (132):
- United States (67):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Encinitas, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, North Hollywood, California
  - Research Site, Orange, California
  - Research Site, Palmdale, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Santa Monica, California
  - Research Site, Stockton, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lynn Haven, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Paducah, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Plymouth, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Ocean City, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Lake Oswego, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Upland, Pennsylvania
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Clinton, Utah
  - Research Site, Bellingham, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (2):
  - Research Site, New Lambton, New South Wales
  - Research Site, Nedlands, Western Australia
- Canada (10):
  - Research Site, Sherwood Park, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Brampton, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Trois-Rivières, Quebec
- France (7):
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Pessac
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Tours
- Germany (9):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cottbus
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, Radebeul
  - Research Site, Rüdersdorf
- Greece (5):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Chaidari, Athens
  - Research Site, Heraklion - Crete
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Ireland (2):
  - Research Site, Cork
  - Research Site, Dublin
- Italy (8):
  - Research Site, Catania
  - Research Site, Ferrara
  - Research Site, Genova
  - Research Site, Modena
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Tradate (VA)
- New Zealand (3):
  - Research Site, Christchurch
  - Research Site, Dunedin
  - Research Site, Remuera
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Skierniewice
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Zgierz
- Research Site, San Juan, Puerto Rico
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (4):
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Wonju-si, Gangwon-do
- Research Site, Taipei, Taiwan

REFERENCES:
- [Background] Globe G, Wiklund I, Mattera M, Zhang H, Revicki DA. Evaluating minimal important differences and responder definitions for the asthma symptom diary in patients with moderate to severe asthma. J Patient Rep Outcomes. 2019 Apr 3;3(1):22. doi: 10.1186/s41687-019-0109-2. PMID 30945020
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 157 centers in Asia, Australia, Canada, Europe, and the United States.
Pre-assignment Details: Participants underwent 3 run-in visits over 4 weeks after completing screening assessments and meeting eligibility criteria. After the run-in visits, eligibility of asthma control questionnaire (ACQ), forced expiratory volume in 1 second (FEV1), and reversibility were confirmed. Eligible participants were randomized in a 1:1 ratio to 1 of 2 arms, stratified based on the current use of long acting β-agonist (LABAs) and number of prior exacerbations (≤ 2 or > 2) in the past year before screening.
Groups:
- Placebo: Participants received placebo subcutaneous injections on day 1 and weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 22.
- Brodalumab 210 mg: Participants received brodalumab 210 mg administered by subcutaneous injection on day 1 and weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 22.
Period: Overall Study
Arm/Group | Placebo | Brodalumab 210 mg
Started | 210 | 211
Received Study Drug | 207 | 208
Completed (Completed end of study visit at week 28) | 162 | 158
Not Completed | 48 | 53
Not completed — Withdrawal by Subject | 19 | 27
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 1 | 0
Not completed — Sponsor Decision | 26 | 24

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Brodalumab 210 mg | Total
Number analyzed (Participants) | 207 | 208 | 415
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.3) | 47.2 (14.0) | 47.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 122 | 242
  Male | 87 | 86 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 21
  Not Hispanic or Latino | 199 | 195 | 394
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 13 | 23
  Black or African American | 29 | 19 | 48
  Multiple | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 162 | 174 | 336
  Other | 3 | 0 | 3
Randomization Strata [Count of Participants; unit: Participants] — Data reported are corrected for errors entered into the Interactive Voice Response System (IVRS) at randomization.
  Participants
    LABA -No; ≤ 2 asthma exacerbation prior year | 30 | 37 | 67
    LABA -No; > 2 asthma exacerbation prior year | 0 | 1 | 1
    LABA -Yes; ≤ 2 asthma exacerbation prior year | 160 | 153 | 313
    LABA -Yes; > 2 asthma exacerbation prior year | 17 | 17 | 34
Duration of Asthma [Mean (Standard Deviation); unit: years] | 22.20 (14.89) | 22.92 (14.44) | 22.56 (14.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Composite Score at Week 24
Description: The ACQ is a validated instrument used in clinical research and practice to evaluate asthma control/impairment.
  The ACQ assesses disease control by evaluating 7 questions: night time awakenings, asthma symptoms upon wakening, activity limitation, shortness of breath, wheeze frequency, short-acting bronchodilator use, and FEV1. All seven items are scored on a 7-point scale, with 0 indicating good control and 6 indicating poor control; the total score is the mean of the seven items and ranges from 0 (totally-controlled) to 6 (extremely poorly controlled). A negative change from baseline indicates improvement. A change of 0.50 points is considered clinically meaningful and a total score of < 1.0 indicates good asthma control.
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 147 | 137
score on a scale | -0.815 (0.073) | -0.865 (0.074)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.5219, Mixed-effect model; The model included fixed effects of treatment group, time, interaction of treatment group by time, stratification variables, and baseline ACQ score; Difference = -0.050, 95% CI 2-sided [-0.203 to 0.103] — Difference = Brodalumab - Placebo

2. Secondary Outcome: Asthma Exacerbation Rate
Description: The asthma exacerbation event rate is defined as the number of events per subject-year during the 24 week treatment period. An asthma exacerbation was defined as an asthma worsening that requires systemic corticosteroids for at least 3 days during the study; distinct asthma exacerbations were defined as events with start dates more than 10 days apart from each other.
Time Frame: Baseline to week 24
Population: Full analysis set with available data
Measure: Number; unit: exacerbations per subject-year
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 204 | 205
exacerbations per subject-year | 0.57 | 0.81
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.102, Generalized linear model; Generalized linear model under a negative binomial distribution assumption adjusting for stratification factors; Rate Ratio = 1.41, 95% CI 2-sided [0.93 to 2.12] — Rate ratio = Brodalumab : Placebo

3. Secondary Outcome: Change From Baseline in ACQ Composite Score at Week 24 in ICS+LABA Subpopulation
Description: as for outcome 1
Time Frame: Baseline and week 24
Population: Full analysis set participants who were taking both inhaled corticosteroids (ICS) and a long-acting β-agonist (LABA) at baseline with available data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 121 | 108
score on a scale | -0.793 (0.084) | -0.831 (0.088)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.6632, Mixed-effect model; The model included fixed effects of treatment group, time, interaction of treatment group by time, stratification factors, and baseline ACQ score; Difference = -0.038, 95% CI 2-sided [-0.210 to 0.134] — Difference = Brodalumab - Placebo

4. Secondary Outcome: Asthma Exacerbation Rate in ICS+LABA Subpopulation
Description: as for outcome 2
Time Frame: Baseline to week 24
Population: Full analysis set participants taking both ICS and LABA at baseline with available data
Measure: Number; unit: exacerbations per subject-year
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 174 | 167
exacerbations per subject-year | 0.60 | 0.89
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.096, Generalized linear model; Generalized linear model under a negative binomial distribution assumption adjusting for stratification factors; Rate Ratio = 1.45, 95% CI 2-sided [0.94 to 2.24] — Rate ratio = Brodalumab : Placebo

5. Secondary Outcome: Change From Baseline in Daily Asthma Symptom Score (7-day Average Score)
Description: The Asthma Symptom Diary (ASD) consists of 23 questions answered on a handheld device, including 10 asthma symptom-related items (5 answered in the morning and 5 in the evening).
  The morning diary comprises questions on 4 asthma-related symptoms (wheezing, shortness of breath, cough, chest tightness), rated on a 5-point severity scale from 0 (no symptom) to 4 (very severe symptoms), and 1 question on nocturnal awakenings, rated from 0 (did not wake up) to 4 (unable to sleep due to asthma). The evening diary has questions on the same 4 asthma-related symptoms and 1 question on limitations of activities, rated from 0 (not at all) to 4 (extremely).
  The ASD daily score is computed by averaging the responses to the 10 symptom-related items, and the mean 7-day ASD score is calculated by averaging the 7 daily scores, with the final score ranging from 0 (minimal symptoms) to 4 (very severe symptoms).
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 121 | 117
score on a scale | -0.397 (0.042) | -0.443 (0.043)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.3290, Mixed-effect model; The model included fixed effects of treatment group, time, interaction of treatment group by time, stratification variables, and baseline score; Difference = -0.046, 95% CI 2-sided [-0.137 to 0.046] — Difference = Brodalumab - Placebo

6. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: L/s
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 148 | 137
L/s | 0.207 (0.045) | 0.237 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.4549, Mixed-effect model; Model includes treatment, time, stratification factors, treatment by time and baseline value of age, gender, pooled race group, height and FEV1; Difference = 0.030, 95% CI [-0.049 to 0.109] — Difference = Brodalumab - Placebo

7. Secondary Outcome: Change From Baseline in Daily Rescue Short-acting Beta-agonist Use
Description: Participants were permitted allowed to use their inhaled rescue medication (SABA) as needed throughout the study and the use was captured in the daily electronic diary (eDiary).
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: puffs
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 121 | 117
puffs | -1.359 (0.243) | -1.231 (0.246)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.6317, Mixed-effect model; The model included fixed effects of treatment group, time, interaction of treatment group by time, stratification variables, and baseline value; Difference = 0.128, 95% CI [-0.396 to 0.653] — Difference = Brodalumab - Placebo

8. Secondary Outcome: Time to First Asthma Exacerbation
Description: An asthma exacerbation is defined as an asthma worsening that requires systemic corticosteroids for at least 3 days during the study. Median time to first asthma exacerbation could not be estimated, the percentage of participants with an asthma exacerbation is reported.
Time Frame: From first dose of study drug to week 24
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 204 | 205
percentage of participants | 20.1 | 23.9
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.238, Log Rank; Log rank test stratified for baseline stratification factors; Hazard Ratio (HR) = 1.277, 95% CI 2-sided [0.843 to 1.936]

9. Secondary Outcome: Number of Participants Who Experienced an Asthma Exacerbation
Description: An asthma exacerbation is defined as an asthma worsening that requires systemic corticosteroids for at least 3 days during the study.
Time Frame: Baseline to week 24
Population: Full analysis set with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 204 | 205
Participants | 41 | 49
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.351, Regression, Logistic; Logistic regression adjusted for stratification factors; Odds Ratio (OR) = 1.25, 95% CI [0.78 to 2.01]

10. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Overall Score
Description: The AQLQ is an asthma-specific instrument that includes evaluations of both symptoms and health-related quality of life measures. The 32-item instrument measures 4 domains affected by asthma including activity limitations, emotional function, exposure to environmental stimuli, and symptoms.
  Participants were asked to recall their experiences during the last 2 weeks and to respond to each question on a 7-point scale (7=no impairment, 1=severe impairment). The overall score was calculated as mean of the responses to the 32 questions and ranges from 1 (severe impairment) to 7 (no impairment). A positive change from baseline indicates improvement.
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 147 | 137
score on a scale | 0.804 (0.085) | 0.803 (0.087)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.9870, Mixed-effects model; The model included fixed effects of treatment group, time, interaction of treatment group by time, stratification variables, and baseline AQLQ score; Difference = -0.001, 95% CI [-0.174 to 0.171] — Difference = Brodalumab - Placebo

11. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow Rate (PEFR)
Description: Peak expiratory flow rate was measured by the participant twice daily at approximately the same time each day (eg, within 1 hour of waking and immediately before bedtime) using a peak flow meter.
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 146 | 129
L/min
  Morning peak flow | 0.072 (5.813) | 0.706 (5.885)
  Evening peak flow: number analyzed (Participants) | 135 | 129
  Evening peak flow | -10.008 (5.719) | -4.089 (5.771)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Analysis of morning peak flow; Test type: Superiority; p = 0.9053, Mixed-effect model; Model includes treatment, time, stratification factors, treatment by time and baseline value of age, gender, pooled race group, height and AM PEFR; Difference = 0.635, 95% CI 2-sided [-9.820 to 11.089] — Difference = Brodalumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Brodalumab 210 mg; Analysis of evening peak flow; Test type: Superiority; p = 0.2661, Mixed-effects model; Model includes treatment, time, stratification factors, treatment by time and baseline value of age, gender, pooled race group, height and PM PEFR; Difference = 5.920, 95% CI 2-sided [-4.515 to 16.354] — Difference = Brodalumab - Placebo

12. Secondary Outcome: Change From Baseline in Variation of Peak Flow
Description: Peak flow was measured by the participant twice daily at approximately the same time each day (eg, within 1 hour of waking and immediately before bedtime) using a peak flow meter. The variation of peak flow is defined as the absolute value of the difference between the A.M. and P.M. peak flow in one day for an individual participant.
Time Frame: Baseline and week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 121 | 115
L/min | -0.872 (2.135) | -4.892 (2.169)
Statistical Analysis 1: Comparison: Placebo vs Brodalumab 210 mg; Test type: Superiority; p = 0.0871, Mixed-effect model; Model includes treatment, time, stratification factors, treatment by time and baseline value of age, gender, race group, height and PEFR variation; Difference = -4.021, 95% CI 2-sided [-8.627 to 0.586] — Difference = Brodalumab - Placebo

13. Secondary Outcome: Proportion of Asthma Symptom-free Days in 4-weeks Intervals Over the Treatment Period
Description: Asthma symptom-free days is defined as days that a participant had a score of zero in their daily asthma symptom diary score.
  The ASD consists of 23 questions answered on a handheld device, including 10 asthma symptom-related items (5 answered in the morning and 5 in the evening).
  The morning diary comprises questions on 4 asthma-related symptoms (wheezing, shortness of breath, cough, chest tightness), rated on a 5-point severity scale from 0 (no symptom) to 4 (very severe symptoms), and 1 question on nocturnal awakenings, rated from 0 (did not wake up) to 4 (unable to sleep due to asthma). The evening diary has questions on the same 4 asthma-related symptoms and 1 question on limitations of activities, rated from 0 (not at all) to 4 (extremely).
  The daily score is the average of the responses to the 10 items.
Time Frame: Baseline (the 4 weeks prior to first dose) and 4-week intervals up to week 24
Population: Full analysis set with available data during each 4-week interval
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 204 | 205
proportion of days
  Baseline: number analyzed (Participants) | 204 | 203
  Baseline | 0.071 (0.179) | 0.041 (0.125)
  Week 4: number analyzed (Participants) | 204 | 203
  Week 4 | 0.122 (0.239) | 0.083 (0.195)
  Week 8: number analyzed (Participants) | 193 | 192
  Week 8 | 0.174 (0.302) | 0.132 (0.268)
  Week 12: number analyzed (Participants) | 185 | 184
  Week 12 | 0.191 (0.319) | 0.164 (0.298)
  Week 16: number analyzed (Participants) | 176 | 174
  Week 16 | 0.211 (0.328) | 0.194 (0.335)
  Week 20: number analyzed (Participants) | 167 | 162
  Week 20 | 0.222 (0.346) | 0.203 (0.339)
  Week 24: number analyzed (Participants) | 160 | 153
  Week 24 | 0.237 (0.371) | 0.204 (0.342)

14. Secondary Outcome: Serum Brodalumab Concentration
Description: Serum brodalumab concentrations were measured using an enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) = 0.0500 µg/mL; values below the LLOQ were set to zero.
Time Frame: Day 1 and weeks 1, 2, 4, 8, 12, 16, and 22 at predose, week 2 + 3 days, week 22 + 3, 7, 10, and 14 days
Population: Participants who received brodalumab with available concentration data at each time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Brodalumab 210 mg
Number analyzed (Participants) | 196
µg/mL
  Day 1 predose | 0 (0)
  Week 1 predose | 8.48 (5.55)
  Week 2 predose: number analyzed (Participants) | 178
  Week 2 predose | 16.8 (9.85)
  Week 2 day 3: number analyzed (Participants) | 50
  Week 2 day 3 | 24.9 (15.8)
  Week 4 predose: number analyzed (Participants) | 174
  Week 4 predose | 14.5 (9.28)
  Week 8 predose: number analyzed (Participants) | 174
  Week 8 predose | 11.1 (9.03)
  Week 12 predose: number analyzed (Participants) | 161
  Week 12 predose | 10.6 (9.86)
  Week 16 predose: number analyzed (Participants) | 150
  Week 16 predose | 8.93 (9.06)
  Week 22 predose: number analyzed (Participants) | 136
  Week 22 predose | 8.94 (9.32)
  Week 22 day 3: number analyzed (Participants) | 46
  Week 22 day 3 | 18.0 (15.4)
  Week 22 day 7: number analyzed (Participants) | 46
  Week 22 day 7 | 14.8 (13.3)
  Week 22 day 10: number analyzed (Participants) | 43
  Week 22 day 10 | 12.5 (12.2)
  Week 22 day 14: number analyzed (Participants) | 146
  Week 22 day 14 | 9.06 (9.78)

15. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.
  The investigator assessed whether the adverse event was possibly related to the investigational product.
  A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal;
  * life threatening;
  * requires in-patient hospitalization or prolongation of existing hospitalization;
  * results in persistent or significant disability/incapacity;
  * congenital anomaly/birth defect;
  * other medically important serious event.
Time Frame: From first dose of study drug up to the end of study, 28 weeks
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brodalumab 210 mg
Number analyzed (Participants) | 207 | 208
Participants
  Any treatment-emergent adverse event | 134 | 156
  TEAE ≥ 2 | 97 | 103
  Serious adverse events | 8 | 7
  TEAE leading to discontinuation of study drug | 9 | 13
  Life-threatening adverse events | 2 | 1
  Fatal adverse events | 1 | 0
  Treatment-related treatment-emergent adverse events | 27 | 44
  Treatment-related TEAE ≥ 2 | 17 | 14
  Treatment-related serious adverse events | 4 | 0
  Treatment-related TEAE leading to discontinuation of study drug | 5 | 8
  Treatment-related life-threatening adverse events | 1 | 0
  Treatment related fatal adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until the end of study, week 28.
Arm/Group | Placebo | Brodalumab 210 mg
Serious Adverse Events (participants affected / at risk) | 8/207 | 7/208
Other Adverse Events (participants affected / at risk) | 104/207 | 129/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=207) | Brodalumab 210 mg (N=208)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=207) | Brodalumab 210 mg (N=208)
Nausea (Gastrointestinal disorders) | 3 | 6
Fatigue (General disorders) | 5 | 2
Injection site erythema (General disorders) | 3 | 6
Bronchitis (Infections and infestations) | 14 | 13
Influenza (Infections and infestations) | 1 | 8
Nasopharyngitis (Infections and infestations) | 19 | 24
Sinusitis (Infections and infestations) | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 19 | 24
Viral upper respiratory tract infection (Infections and infestations) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Headache (Nervous system disorders) | 11 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 63 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.